CLINICAL TRIAL: NCT04851691
Title: A Pragmatic Randomized-controlled Trial of a Multi-pronged Electronic Health Record-based Clinical Decision Support Tool to Reduce Low-value Antipsychotic Prescriptions Among Older Adults With Alzheimer's and Related Dementias
Brief Title: An Electronic Clinical Decision Support Tool to Reduce Low-value Antipsychotic Prescriptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Catherine A. Sarkisian, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01AG059815-01S1 (NIH); 1R01AG059815-01 (NIH); R01AG059815-01S1 (NIH)
Record Dates: First submitted 2021-04-02; First posted 2021-04-20 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease; Dementia Alzheimers; Dementia of Alzheimer Type
Keywords: Low Value Care; Antipsychotic medication
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EHR CDS tool (Experimental): Patients with an encounter in which the physician attempts to place an order for a new antipsychotic prescription. Physician has been assigned to the EHR CDS tool.
  Multi-pronged electronic health record (EHR) clinical decision support (CDS) tool intervention to reduce physician prescriptions of new antipsychotic medications among older adults with ADRD
  Interventions: Behavioral: EHR CDS
- Control (Experimental): Patients with an encounter in which the physician attempts to place an order for a new antipsychotic prescription. Physician has been assigned to the control.
  Physicians will not receive intervention and perform duties as usual.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: EHR CDS — When a clinician initiates a new antipsychotic prescription for a patient with dementia, a three-pronged electronic health record clinical decision support tool "pops up": (1) Alerting clinicians that antipsychotic prescriptions increase patient mortality; (2) Offering non-pharmacological behavioral resources for caregivers via a link to the IDEA! strategy resources on how caregivers can best manage a patient's behavioral disturbance non-pharmacologically, which will be available in the EHR to include in the patient's after visit summary; and (3) Defaulting prescriptions to a low supply of pills in to order to minimize harm. In addition, the PI will email all providers randomized to the intervention arm in order to make them aware of the components of this intervention and its motivation.
  Arms: EHR CDS tool
Other: Usual Care — Patients will receive usual care from their physicians.
  Arms: Control

SUMMARY:
The goal of this study will be to design, implement and test the impact of a quality improvement (QI) intervention that uses an EHR CDS tool among physicians newly ordering an antipsychotic medication for older adults with ADRD. The study team hypothesizes that the intervention will reduce each participating clinician's pill days per patient prescribed.

DETAILED DESCRIPTION:
Importance: Among patients with Alzheimer's disease and its related dementias (ADRD) with behavioral disturbances, antipsychotic prescriptions have limited efficacy and substantially increase risk of death. Despite an FDA 2005 "black box" warning and multiple professional physician society guidelines discouraging their use, physicians continue to frequently prescribe antipsychotic medications as first-line therapy for behavioral disturbances among patients with ADRD.

Objective: This study will measure the impact of a multi-pronged electronic health record (EHR) clinical decision support (CDS) tool intervention to reduce physician prescriptions of new antipsychotic medications among older adults with ADRD.

Design, Setting, and Participants: Utilizing a pragmatic parallel cluster-randomized trial design, the study will randomize eligible physicians from a large urban academic medical center to either receive an EHR CDS tool (intervention) or not (control) when they prescribe a new antipsychotic medication during a visit with a patient with ADRD. The intervention will include three components: (1) alerts the prescriber that antipsychotic prescriptions increase mortality; (2) offers non-pharmacological behavioral resources for caregivers; and if the prescriber does not cancel the order (3) auto-defaults the prescription to contain the lowest dose and number of pills (n=30) without refills. In addition, the PI will email all providers randomized to the intervention arm in order to make them aware of the components of this intervention and its motivation. Acknowledging the clinical complexity of this vulnerable patient population, the multidisciplinary study team attempted to design the intervention to maximize impact while minimizing clinician burden. Over a one-year timeframe, the study team will compare the cumulative total of new antipsychotic pill-days prescribed (primary outcome) by physicians in the intervention group versus in the control group.

Hypothesis: This pragmatic trial will advance understanding of how a multi-pronged EHR CDS tool can potentially reduce harmful, low-value care among older adults with ADRD.

ELIGIBILITY:
Inclusion Criteria:

* Physicians who will be eligible to receive the EHR CDS tool intervention include those who provide ambulatory care in the UCLA health system and have newly prescribed antipsychotics (e.g., Quetiepine, Olanzapine, Risperidone, Aripiprazole, Haloperidol, Clozapine) for eligible patients (described below) at the medical center in the last 24 months.
* Eligible patients will be enrolled in the study during their first encounter with one of the randomized physicians (see above) during which a new antipsychotic medication order will be initiated. Inclusion criteria for patients will include: 1) having an assigned primary care physician (PCP) and/or assignment to an Accountable Care Organization (ACO) at UCLA Health, and: 2) being part of the health system's EHR-based dementia registry.

Exclusion Criteria:

* Patients who have diagnosis codes for schizophrenic disorders, delusion disorders, bipolar disorders, or other non-organic psychoses on their problem list.
* Patients with Parkinson's disease on their problem list
* Patients who have been prescribed antipsychotics in the prior 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Sarkisian, MD, MSPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Health, Los Angeles, California, United States

REFERENCES:
- [Background] Schneider LS, Tariot PN, Dagerman KS, Davis SM, Hsiao JK, Ismail MS, Lebowitz BD, Lyketsos CG, Ryan JM, Stroup TS, Sultzer DL, Weintraub D, Lieberman JA; CATIE-AD Study Group. Effectiveness of atypical antipsychotic drugs in patients with Alzheimer's disease. N Engl J Med. 2006 Oct 12;355(15):1525-38. doi: 10.1056/NEJMoa061240. PMID 17035647
- [Background] Hwang YJ, Dixon SN, Reiss JP, Wald R, Parikh CR, Gandhi S, Shariff SZ, Pannu N, Nash DM, Rehman F, Garg AX. Atypical antipsychotic drugs and the risk for acute kidney injury and other adverse outcomes in older adults: a population-based cohort study. Ann Intern Med. 2014 Aug 19;161(4):242-8. doi: 10.7326/M13-2796. PMID 25133360
- [Background] Maher AR, Maglione M, Bagley S, Suttorp M, Hu JH, Ewing B, Wang Z, Timmer M, Sultzer D, Shekelle PG. Efficacy and comparative effectiveness of atypical antipsychotic medications for off-label uses in adults: a systematic review and meta-analysis. JAMA. 2011 Sep 28;306(12):1359-69. doi: 10.1001/jama.2011.1360. PMID 21954480
- [Background] American Geriatrics Society. Ten things clinicians and patients should question. Choosing wisely: an initiative of the ABIM foundation. http://www.choosingwisely.org/societies/american-geriatrics-society/. Accessed Revised April 23, 2015.
- [Background] Reus VI, Fochtmann LJ, Eyler AE, Hilty DM, Horvitz-Lennon M, Jibson MD, Lopez OL, Mahoney J, Pasic J, Tan ZS, Wills CD, Rhoads R, Yager J. The American Psychiatric Association Practice Guideline on the Use of Antipsychotics to Treat Agitation or Psychosis in Patients With Dementia. Am J Psychiatry. 2016 May 1;173(5):543-6. doi: 10.1176/appi.ajp.2015.173501. No abstract available. PMID 27133416
- [Background] Kuehn BM. FDA warns antipsychotic drugs may be risky for elderly. JAMA. 2005 May 25;293(20):2462. doi: 10.1001/jama.293.20.2462. No abstract available. PMID 15914734
- [Background] Maust DT, Strominger J, Bynum JPW, Langa KM, Gerlach LB, Zivin K, Marcus SC. Prevalence of Psychotropic and Opioid Prescription Fills Among Community-Dwelling Older Adults With Dementia in the US. JAMA. 2020 Aug 18;324(7):706-708. doi: 10.1001/jama.2020.8519. PMID 32808997
- [Background] Morgan DJ, Leppin AL, Smith CD, Korenstein D. A Practical Framework for Understanding and Reducing Medical Overuse: Conceptualizing Overuse Through the Patient-Clinician Interaction. J Hosp Med. 2017 May;12(5):346-351. doi: 10.12788/jhm.2738. PMID 28459906
- [Background] Colla CH. Swimming against the current--what might work to reduce low-value care? N Engl J Med. 2014 Oct 2;371(14):1280-3. doi: 10.1056/NEJMp1404503. No abstract available. PMID 25271601
- [Background] Mafi JN, Parchman M. Low-value care: an intractable global problem with no quick fix. BMJ Qual Saf. 2018 May;27(5):333-336. doi: 10.1136/bmjqs-2017-007477. Epub 2018 Jan 13. No abstract available. PMID 29331955
- [Background] Bourdeaux CP, Davies KJ, Thomas MJ, Bewley JS, Gould TH. Using 'nudge' principles for order set design: a before and after evaluation of an electronic prescribing template in critical care. BMJ Qual Saf. 2014 May;23(5):382-8. doi: 10.1136/bmjqs-2013-002395. Epub 2013 Nov 26. PMID 24282310
- [Background] Davidai S, Gilovich T, Ross LD. The meaning of default options for potential organ donors. Proc Natl Acad Sci U S A. 2012 Sep 18;109(38):15201-5. doi: 10.1073/pnas.1211695109. Epub 2012 Sep 4. PMID 22949639
- [Background] Patel MS, Day SC, Halpern SD, Hanson CW, Martinez JR, Honeywell S Jr, Volpp KG. Generic Medication Prescription Rates After Health System-Wide Redesign of Default Options Within the Electronic Health Record. JAMA Intern Med. 2016 Jun 1;176(6):847-8. doi: 10.1001/jamainternmed.2016.1691. No abstract available. PMID 27159011
- [Background] Sacarny A, Barnett ML, Le J, Tetkoski F, Yokum D, Agrawal S. Effect of Peer Comparison Letters for High-Volume Primary Care Prescribers of Quetiapine in Older and Disabled Adults: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Oct 1;75(10):1003-1011. doi: 10.1001/jamapsychiatry.2018.1867. PMID 30073273
- [Background] Roddy E, Jones E. On Hippocrates. Hippocratic ideals are alive and well in 21st century. BMJ. 2002 Aug 31;325(7362):496. doi: 10.1136/bmj.325.7362.496/a. No abstract available. PMID 12202343
- [Background] Liao JM, Schapira MS, Navathe AS, Mitra N, Weissman A, Asch DA. The Effect of Emphasizing Patient, Societal, and Institutional Harms of Inappropriate Antibiotic Prescribing on Physician Support of Financial Penalties: A Randomized Trial. Ann Intern Med. 2017 Aug 1;167(3):215-216. doi: 10.7326/L17-0102. Epub 2017 Jun 20. No abstract available. PMID 28631001
- [Background] Schpero WL, Morden NE, Sequist TD, Rosenthal MB, Gottlieb DJ, Colla CH. For Selected Services, Blacks And Hispanics More Likely To Receive Low-Value Care Than Whites. Health Aff (Millwood). 2017 Jun 1;36(6):1065-1069. doi: 10.1377/hlthaff.2016.1416. PMID 28583965
- [Background] Seppi K, Ray Chaudhuri K, Coelho M, Fox SH, Katzenschlager R, Perez Lloret S, Weintraub D, Sampaio C; the collaborators of the Parkinson's Disease Update on Non-Motor Symptoms Study Group on behalf of the Movement Disorders Society Evidence-Based Medicine Committee. Update on treatments for nonmotor symptoms of Parkinson's disease-an evidence-based medicine review. Mov Disord. 2019 Feb;34(2):180-198. doi: 10.1002/mds.27602. Epub 2019 Jan 17. PMID 30653247
- [Background] Colla CH, Morden NE, Sequist TD, Schpero WL, Rosenthal MB. Choosing wisely: prevalence and correlates of low-value health care services in the United States. J Gen Intern Med. 2015 Feb;30(2):221-8. doi: 10.1007/s11606-014-3070-z. Epub 2014 Nov 6. PMID 25373832

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were enrolled into the study when an eligible provider initiated a new antipsychotic prescription (e.g., Quetiapine, Olanzapine, Risperidone, Aripiprazole, Haloperidol, Clozapine) during a patient visit. Eligible providers were assigned an arm of the study based on their 2019 new antipsychotic orders for this population. Patients were enrolled into each arm based on the providers arm assignment. Healthcare Providers were not enrolled in the study.
Groups:
- EHR CDS Tool: Patients with an encounter in which the physician attempts to place an order for a new antipsychotic prescription. Physician has been assigned to the EHR CDS tool.
  The three-pronged electronic health record clinical decision support tool "pops up": (1) Alerting clinicians that antipsychotic prescriptions increase patient mortality; (2) Offering non-pharmacological behavioral resources for caregivers via a link to the IDEA! strategy resources on how caregivers can best manage a patient's behavioral disturbance non-pharmacologically, which will be available in the EHR to include in the patient's after visit summary; and (3) Defaulting prescriptions to a low supply of pills in to order to minimize harm. In addition, the PI will email all providers randomized to the intervention arm in order to make them aware of the components of this intervention and its motivation.
- Control: Patients with an encounter in which the physician attempts to place an order for a new antipsychotic prescription. Physician has been assigned to the control.
  Usual Care: Patients will receive usual care from their physicians.
Period: Overall Study
Arm/Group | EHR CDS Tool | Control
Started | 67 | 91
Completed | 67 | 91
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Providers were not assessed for baseline
Groups:
- EHR CDS Tool: Patients with an encounter in which the physician attempts to place an order for a new antipsychotic prescription. Physician has been assigned to the EHR CDS tool.
  Multi-pronged electronic health record (EHR) clinical decision support (CDS) tool intervention to reduce physician prescriptions of new antipsychotic medications among older adults with ADRD
  EHR CDS: When a clinician initiates a new antipsychotic prescription for a patient with dementia, a three-pronged electronic health record clinical decision support tool "pops up": (1) Alerting clinicians that antipsychotic prescriptions increase patient mortality; (2) Offering non-pharmacological behavioral resources for caregivers via a link to the IDEA! strategy resources on how caregivers can best manage a patient's behavioral disturbance non-pharmacologically, which will be available in the EHR to include in the patient's after visit summary; and (3) Defaulting prescriptions to a low supply of pills in to order to minimize harm. In addition, the PI will email all providers randomized to the intervention arm in order to make them aware of the components of this intervention and its motivation.
- Control: Patients with an encounter in which the physician attempts to place an order for a new antipsychotic prescription. Physician has been assigned to the control.
  Physicians will not receive intervention and perform duties as usual.
  Usual Care: Patients will receive usual care from their physicians.
- Total: Total of all reporting groups
Arm/Group | EHR CDS Tool | Control | Total
Number analyzed (Participants) | 67 | 91 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.19 (15.14) | 84.78 (11.77) | 83.26 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 65 | 106
  Male | 26 | 26 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 70 | 122
  Not Hispanic or Latino | 6 | 10 | 16
  Unknown or Not Reported | 9 | 11 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race Category: Asian | 5 | 7 | 12
  Race Category: Other Race | 3 | 7 | 10
  Race Category: White | 45 | 63 | 108
  Race Category: Unknown or Not Reported | 8 | 11 | 19
  Race Category: Black or African American | 5 | 3 | 8
  Race Category: American Indian or Alaska Native | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Total of New Antipsychotic Pill-days Prescribed
Description: Cumulative total of new antipsychotic prescription days supplied by clinicians per eligible patient in the 12 months after the intervention rollout date compared to the prior 12-months
Time Frame: 12 month time point
Population: Patients that received a new antipsychotic prescription (e.g., Quetiapine, Olanzapine, Risperidone, Aripiprazole, Haloperidol, Clozapine) from an eligible provider.
Measure: Number; unit: New antipsychotic prescription days
Arm/Group | EHR CDS Tool | Control
Number analyzed (Participants) | 67 | 91
New antipsychotic prescription days | 12569 | 25916

2. Secondary Outcome: Number of Patients Who Receive Handout
Description: Number of patients who receive the non-Pharmacologic IDEA Strategy handout at 12 month time point comparing the intervention vs. control
Time Frame: 12 month time point
Population: All participants enrolled in the study were eligible to receive the non-Pharmacologic IDEA Strategy handout
Measure: Count of Participants; unit: Participants
Arm/Group | EHR CDS Tool | Control
Number analyzed (Participants) | 67 | 91
Participants | 0 | 0

3. Secondary Outcome: Number of Patients With ER Visit
Description: Number of patients with at least one emergency department visit within 90 days of being exposed to the intervention
Time Frame: 90 days
Reporting Status: Not Posted

4. Secondary Outcome: Number of Patients With Hospitalization
Description: Number of patients with at least one hospitalization within 90 days of being exposed to the intervention
Time Frame: 90 days
Reporting Status: Not Posted

5. Secondary Outcome: Hospitalizations (Including Psychiatric Hospitalizations)
Description: Hospitalizations (including psychiatric hospitalizations) within 90 days of being exposed to the intervention
Time Frame: 90 days
Reporting Status: Not Posted

6. Secondary Outcome: Death Within 90 Days After Enrollment
Description: Death within 90 days after enrollment
Time Frame: 90 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Participants were tracked for adverse events 3 months after their first encounter with a randomized physician during which a new antipsychotic medication order is initiated.
Description: An adverse event is defined as an Emergency Department visit that did not require hospitalization.
  Serious adverse events include hospitalization or death.
  Providers were not assessed for adverse events
Arm/Group | EHR CDS Tool | Control
All-Cause Mortality (participants affected / at risk) | 1/67 | 2/91
Serious Adverse Events (participants affected / at risk) | 2/67 | 12/91
Other Adverse Events (participants affected / at risk) | 4/67 | 6/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EHR CDS Tool (N=67) | Control (N=91)
Inpatient Admission (General disorders) | 2 | 12 — All cause inpatient admissions of enrolled participants were chart reviewed when admitted up to 30 days following enrollment encounter. All reasons for visit were considered eligible for review
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EHR CDS Tool (N=67) | Control (N=91)
Emergency Department visits that did not require admissions (General disorders) | 4 | 6 — All cause emergency department visits of enrolled participants were chart reviewed when visit occurred up to 30 days following enrollment encounter. All reasons for visit were considered eligible for review

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT04851691/Prot_SAP_000.pdf